CLINICAL TRIAL: NCT04914884
Title: Clinical Application of Intraocular Fluid Detection in Endophthalmitis
Brief Title: Intraocular Fluid Detection in Endophthalmitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Junhui Shen, Dr, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: I2020001874
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Intraocular Inflammation
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intraocular inflammation group
  Interventions: Diagnostic Test: intraocular fluid detection
- Cataract patients group
  Interventions: Diagnostic Test: intraocular fluid detection

INTERVENTIONS:
Diagnostic Test: intraocular fluid detection — This study mainly verified the use of molecular biology technology to detect the changes of VCAM, ICAM-1 and other cytokines, bacteria, viruses, fungi, Toxoplasma gondii IgG in patients' intraocular fluid, including aqueous humor and vitreous humor, so as to timely judge the etiology and progress of endophthalmitis, and provide reference for diagnosis and treatment.

SUMMARY:
Endophthalmitis is also called vitreous inflammation. Broadly speaking, it refers to all kinds of serious intraocular inflammation, such as vitreitis, anterior chamber empyema and eye pain caused by intraocular infection, intraocular foreign body, tumor necrosis, severe non infectious uveitis, lens cortex allergy, etc. Clinically, it generally refers to infectious endophthalmitis caused by bacteria, fungi or parasites. According to the different ways of infection, it can be divided into exogenous endophthalmitis and endogenous endophthalmitis. Exogenous endophthalmitis is more common. When inflammation involves sclera or extraocular orbital tissue, it is called "panophthalmia".

Endophthalmitis is a kind of serious intraocular inflammation which can lead to the loss of visual function. Early diagnosis and treatment is the key. Studies have found that the changes of cytokines in aqueous humor are helpful for the diagnosis of endophthalmitis. Okhrvai et al. Also pointed out that the application of PCR can reduce the diagnosis time of endophthalmitis. This study mainly verified the use of molecular biology technology to detect the changes of VCAM, ICAM-1 and other cytokines, bacteria, viruses, fungi, Toxoplasma gondii IgG in patients' intraocular fluid, including aqueous humor and vitreous humor, so as to timely judge the etiology and progress of endophthalmitis, and provide reference for diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* ① Clinical manifestations: eye pain, photophobia and tears, decreased vision, conjunctival congestion and edema, etc. ② Special examination: anterior examination showed conjunctival congestion and edema, postkeratosis, anterior chamber empyema and other inflammatory manifestations. Fundus examination showed vitreous opacity, fundus hemorrhage and white lesions. ③ Laboratory examination: bacteria, viruses, fungi and Toxoplasma gondii were detected in the aqueous humor and vitreous humor of the patients.

Exclusion Criteria:

* 1. With tumor, rheumatoid and other autoimmune diseases. 2. Accompanied by diabetes and other systemic chronic diseases. 3. Patients with retinal and choroidal vascular diseases and history of eye surgery were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the formula n = Z2 * (p * (1-p)) / E2, the confidence is 95%, the error is 10%, and the probability is 0.5. The sample size is calculated to be 96 cases. According to some similar literatures, the sample size is set to be 100 cases.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The intraocular fluid of patients with endophthalmitis and age-related cataract were collected | 2021.1-2021.6
  to check the cytokines in the intraocular fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No